CLINICAL TRIAL: NCT04918225
Title: Motor Asymmetry in Progressive Multiple Sclerosis Patients
Acronym: MAP-MS
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_9751_MAP-MS
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
Keywords: motor disability, Magnetic Resonance Imaging
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Magnetic Resonance Spectroscopy; Neurologic Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Progressive Multiple Sclerosis patients: Progressive Multiple Sclerosis patients
  Interventions: Radiation: Magnetic Resonance Imaging; Diagnostic Test: Neurological examination; Diagnostic Test: Multiple Sclerosis Functional Composite; Diagnostic Test: Physiotherapist examination
- Healthy Volunteers: Healthy Volunteers
  Interventions: Radiation: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging — Encephalic (about 30 minutes*)
  * lesion location assessment: 3D FLAIR, 3DT1, 3DT2 (standard OFSEP protocol)
  * lesion severity assessment: Axial magnetization transfer imaging (mt0, mt1)
  * tract location assessment: 30 directions diffusion imaging (standard OFSEP protocol)
  * B0 and B1 mapping to correct for B0 and B1 inhomogeneities
    ● Spinal cord (about 50 minutes*)
  * lesion location assessment: cervical and thoracic sagittal T2 TSE (0.7x0.7x2.5mm3), axial cervical MEDIC T2* (0.7x0.7x3mm3), axial thoracic T2 (0.5x0.5x3mm3)
  * lesion severity assessment: Axial magnetization transfer imaging (mt0, mt1, 0.7x0.7x3mm3) on the cervical cord and on the thoracic cord
  * tract location assessment: performed from registration on atlas
  * B0 and B1 mapping to correct for B0 and B1 inhomogeneities
Diagnostic Test: Neurological examination — Global disability will be scored using the Expanded Disability Status Scale score
  Groups: Progressive Multiple Sclerosis patients
Diagnostic Test: Multiple Sclerosis Functional Composite — * Walking disability will be scored using the 25-foot timed-walked test
  * Arm disability will be scored using the nine-hole peg test
  Groups: Progressive Multiple Sclerosis patients
Diagnostic Test: Physiotherapist examination — * American Society Injury. Association motor subscore for each limb
  * The muscle strength using a dynamometer. Two muscle groups will be tested for the upper (elbow flexors and extensors) and lower limbs (hip flexors and ankle dorsiflexion).
  * The Ashworth Scale and the Tardieu Scale to assess spasticity.
  * 6 minutes walking test
  * Fatigue Severity Scale
  * MFIS : Modified Fatigue Impact Scale
  Groups: Progressive Multiple Sclerosis patients

SUMMARY:
Project Rational

A better understanding of the causes of physical disability is an important unmet need in progressive Multiple Sclerosis patients. Progressive Multiple Sclerosis patients most often present a worsening pyramidal syndrome of lower and, to a lesser extent, upper limbs (Lublin et al., 2014) suggesting a strong corticospinal tract involvement. The systematic high resolution Magnetic Resonance Imaging exploration of lesions location and severity, as well as extra-lesional tissue, on pan-medullar and encephalic motor tracts offers the opportunity to better understand the pathological mechanism associated with motor impairment.

Scientific aims

This project will follow a twofold approach. First, the investigators will consider an "inter-patient" approach where independent and absolute Magnetic Resonance metrics for each limb will be related to disability. Second, the investigators will consider an "intra-patient" approach (i.e. comparing differences of Magnetic Resonance metric and of clinical score from the left and the right side in the same patient). For this purpose, progressive Multiple Sclerosis patients with asymmetric motor impairment will be studied. Confronting clinical and Magnetic Resonance Imaging metric value asymmetries indeed offers the unique opportunity to free oneself from many confounding factors such as genetics, age, duration of disease evolution, acquisition bias, etc. These two approaches will allow us to precisely study the impact of local factors such as Multiple Sclerosis lesions located on motor tracts on motor disability.

Methodology

The investigators propose an observational multicenter cross-sectional and prognostic study. This study will involve two French centers (Rennes, Marseille) and will include a total of 40 progressive Multiple Sclerosis patients with an asymmetrical motor deficit. Twenty sex and age matched controls will be needed to calibrate quantitative Magnetic Resonance imaging (magnetization transfer ratio). Encephalic and pan medullar structural and quantitative Magnetic Resonance images will be acquired at inclusion and clinical follow-up examinations will be performed at inclusion and 24 months. Detailed motor evaluation "per limb" will be performed, including the motor American Society Injury. Association sub-score and upper and lower limbs muscle strength measurements using a dynamometer.

ELIGIBILITY:
1. - Inclusion Criteria:

   1.1/ Patients:
   * Aged between 18 and 60 years.
   * Primary Progressive Multiple Sclerosis or Secondary Progressive Multiple Sclerosis as defined by Mac Donald revised criteria in 2017.
   * Expanded Disability Status Scale lower or equal to 8.0, at inclusion.
   * asymmetric motor deficit. The motor deficit asymmetry will be defined by a difference of 3 or more at the American Society Injury. Association motor sub-score per limb between the right lower limb and the left lower limb.
   * No evidence of focal inflammatory activity for at least 3 years (no clinical relapse, no gadolinium enhancement on an Magnetic Resonance Imaging scan and no new T2 lesion)
   * Provided written informed consent according to the Institutional review board approval
   * Affiliated to the French healthcare system.

   1.2 / Controls:
   * Aged between 18 and 60 years, sex and age matched with patients.
   * Provided written informed consent according to the Institutional review board approval
   * Affiliated to the French healthcare system.
2. - Non-inclusion criteria:

2.1 /Patients:

* cerebellar Expanded Disability Status Scale sub score higher than pyramidal Expanded Disability Status Scale sub score.
* Relapse or corticosteroids in the 30 days preceding inclusion.
* Other neurological diseases.
* Lack of ability to understand the Institutional review board consent form.
* Magnetic Resonance contraindications.
* Pregnancy and breastfeeding.
* Major persons subject to legal protection (legal safeguards, guardianship,curatorship), persons deprived of their liberty

2.2 / Controls:

* Personal history of central nervous related disease
* Familial history of Multiple Sclerosis.
* Personal history of spinal cord injury.
* Personal history of spondylotic myelopathy.
* Magnetic Resonance Imaging contraindication.
* Lack of ability to understand the Institutional review board form.
* Major persons subject to legal protection (legal safeguards, guardianship, curatorship), persons deprived of their liberty
* Pregnancy and breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient population will consist of progressive Multiple Sclerosis patients (both Primary Progressive Multiple Sclerosis and Secondary Progressive Multiple Sclerosis), a population for whom a better understanding of the causes of disability is an unmet need.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
link between focal and diffuse damage in motor tract | Baseline
  link between focal and diffuse damage in motor tract per side and it functional consequences per limb assessed clinically at baseline

SECONDARY OUTCOMES:
Link between the asymmetry of functional motor impairment and the asymmetry of structural damage on the motor pathways | Baseline
  To study the link between the asymmetry of functional motor impairment and the asymmetry of structural damage on the motor pathways (intra-patient assessment).
prognostic value of motor tract focal and diffuse damage on clinical scores variations | 24 months
  To study the prognostic value of motor tract focal and diffuse damage on clinical scores variations at 2 years
link between fatigability, fatigue and analytical disorders | 24 months
  To explore fatigability during the 6-minute instrumented walking test (evolution of spatio-temporal parameters: walking speed, step length, cadence; feeling of fatigue) and to study the link between fatigability, fatigue and analytical disorders (strength, spasticity)
link between fatigue and fatigability and the focal and diffuse impairment of the motor pathways | 24 months
  To study the link between fatigue and fatigability and the focal and diffuse impairment of the motor pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kerbrat, MD, Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - Hôpital de la Timone, AP-HM, Marseille
  - CHU de Rennes - Hôpital Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No